CLINICAL TRIAL: NCT06494696
Title: Utilizing 68Ga-PSMA PET/MRI Imaging in Conjunction With mpMRI for Evaluating Prospective Prostate Cancer Risk
Brief Title: 68Ga-PSMA PET/MRI in Conjunction With mpMRI for Evaluating Prospective Prostate Cancer Risk
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 202400643A3
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer
Keywords: Ga-68 PSMA PET/MRI; PI-RADS; Biopsy naive
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Experimental
  Interventions: Diagnostic Test: Ga-68 PSMA PET/MRI

INTERVENTIONS:
Diagnostic Test: Ga-68 PSMA PET/MRI — The participant will undergo a Ga-68 PSMA PET/MRI scan, and then be followed up for 2 years to see if prostate cancer is diagnosed.

SUMMARY:
The goal of this observational study is to learn if Ga-68 PSMA PET/MRI can better diagnose prostate cancer than mpMRI in males between 40 to 85 years old who is naive to prostate biopsy and is suspicious for prostate cancer by elevated PSA or lower urinary tract symptoms. The main questions it aims to answer are:

1. Does PSMA PET/MRI have better PPV and NPV than mpMRI to diagnose prostate cancer?
2. Does lesion location concordance in PSMA PET and MRI effect diagnosis accuracy?

Participants will:

1. Undergo a Ga-68 PSMA PET/MRI scan and keep followed up for 2 years to check if prostate cancer is diagnosed after the scan.
2. Between the follow-up period, visit the clinic once every 6 months for checkups and blood tests.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who indicated MRI of pelvis due to clinical suspicion of prostate cancer based on elevated PSA (4~20 ng/mL), abnormal digital rectal examination or lower urinary tract syndromes.
2. Males aged between 40 and 85 years with a life expectancy greater than two years.
3. Naïve to prostate biopsy in the past.
4. Assessment of daily physical status graded 0 to 2 based on the Eastern Cooperative Oncology Group (ECOG) criteria.
5. Willing to sign the informed consent.

Exclusion Criteria:

1. Unable to tolerate the PET/MRI scan, such as those with claustrophobia, unable to lie still, consciousness unclear, vital sign unstable, or having MRI unsafe metallic implants or devices.
2. With renal impairment (glomerular filtration rate lower than 30 ml/min/1.73 m2), and allergy to medium contrast.
3. High risk to conduct examination after evaluations of PI
4. Patient had previous malignancy history

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who indicated MRI of pelvis due to clinical suspicion of prostate cancer based on elevated PSA (4~20 ng/mL), abnormal digital rectal examination or lower urinary tract syndromes.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
PPV of concordant PET/MRI lesion plus PI-RADS score 4~5 | 2 years after PSMA PET/MRI scan
  Comparing positive predictive values (PPV) of using concordant PET/MRI lesion plus PI-RADS score 4~5 as positive test with PPV of using PI-RADS 4~5 alone as positive test to predict diagnosing prostate cancer within 2 years.
NPV of using negative PET lesion plus PI-RADS score 1~3 | 2 years after PSMA PET/MRI scan
  Comparing negative predictive values (NPV) of using negative PET lesion plus PI-RADS score 1~3 as negative test with NPV of using PI-RADS 1~3 alone as negative test to predict diagnosing prostate cancer within 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Ren Tseng, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital ,Linkou, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eiber M, Weirich G, Holzapfel K, Souvatzoglou M, Haller B, Rauscher I, Beer AJ, Wester HJ, Gschwend J, Schwaiger M, Maurer T. Simultaneous 68Ga-PSMA HBED-CC PET/MRI Improves the Localization of Primary Prostate Cancer. Eur Urol. 2016 Nov;70(5):829-836. doi: 10.1016/j.eururo.2015.12.053. Epub 2016 Jan 18. PMID 26795686
- [Background] Al-Bayati M, Grueneisen J, Lutje S, Sawicki LM, Suntharalingam S, Tschirdewahn S, Forsting M, Rubben H, Herrmann K, Umutlu L, Wetter A. Integrated 68Gallium Labelled Prostate-Specific Membrane Antigen-11 Positron Emission Tomography/Magnetic Resonance Imaging Enhances Discriminatory Power of Multi-Parametric Prostate Magnetic Resonance Imaging. Urol Int. 2018;100(2):164-171. doi: 10.1159/000484695. Epub 2018 Jan 25. PMID 29393268
- [Background] Muehlematter UJ, Burger IA, Becker AS, Schawkat K, Hotker AM, Reiner CS, Muller J, Rupp NJ, Ruschoff JH, Eberli D, Donati OF. Diagnostic Accuracy of Multiparametric MRI versus 68Ga-PSMA-11 PET/MRI for Extracapsular Extension and Seminal Vesicle Invasion in Patients with Prostate Cancer. Radiology. 2019 Nov;293(2):350-358. doi: 10.1148/radiol.2019190687. Epub 2019 Sep 10. PMID 31502937
- [Background] Emmett L, Buteau J, Papa N, Moon D, Thompson J, Roberts MJ, Rasiah K, Pattison DA, Yaxley J, Thomas P, Hutton AC, Agrawal S, Amin A, Blazevski A, Chalasani V, Ho B, Nguyen A, Liu V, Lee J, Sheehan-Dare G, Kooner R, Coughlin G, Chan L, Cusick T, Namdarian B, Kapoor J, Alghazo O, Woo HH, Lawrentschuk N, Murphy D, Hofman MS, Stricker P. The Additive Diagnostic Value of Prostate-specific Membrane Antigen Positron Emission Tomography Computed Tomography to Multiparametric Magnetic Resonance Imaging Triage in the Diagnosis of Prostate Cancer (PRIMARY): A Prospective Multicentre Study. Eur Urol. 2021 Dec;80(6):682-689. doi: 10.1016/j.eururo.2021.08.002. Epub 2021 Aug 28. PMID 34465492
- [Background] Bates A, Miles K. Prostate-specific membrane antigen PET/MRI validation of MR textural analysis for detection of transition zone prostate cancer. Eur Radiol. 2017 Dec;27(12):5290-5298. doi: 10.1007/s00330-017-4877-x. Epub 2017 Jun 12. PMID 28608163
- [Background] Tang W, Tang Y, Qi L, Zhang Y, Tang G, Gao X, Hu S, Cai Y. Benign Prostatic Hyperplasia-Related False-Positive of Prostate-Specific Membrane Antigen-Positron Emission Tomography in the Diagnosis of Prostate Cancer: The Achilles' Heel of Biopsy-Free Radical Prostatectomy? J Urol. 2023 Dec;210(6):845-855. doi: 10.1097/JU.0000000000003680. Epub 2023 Aug 30. PMID 37647549
- [Background] Wong LM, Koschel S, Whish-Wilson T, Farag M, Bolton D, Zargar H, Corcoran N, Lawrentschuk N, Christov A, Thomas L, Perry E, Heinze S, Taubman K, Sutherland T. Investigating PSMA-PET/CT to resolve prostate MRI PIRADS4-5 and negative biopsy discordance. World J Urol. 2023 Feb;41(2):463-469. doi: 10.1007/s00345-022-04243-5. Epub 2023 Jan 5. PMID 36602577